CLINICAL TRIAL: NCT00390975
Title: An Open-label Pilot Trial to Assess the Effect of Tegaserod on Improvement of Gastric Emptying in Patients With Diabetic Gastroparesis and Upper Gastrointestinal Symptoms
Brief Title: Effect of Tegaserod on Gastric Emptying in Patients With Diabetic Gastroparesis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was terminated early as a result of regulatory action suspending tegaserod use in 2007
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919GUS62
Record Dates: First submitted 2006-10-20; First posted 2006-10-23 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Gastroparesis; Diabetes
Keywords: Tegaserod; diabetes; diabetic gastroparesis; gastric emptying; gastric retention; electrogastrography
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus | interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
This study will assess gastric emptying in patients with symptoms of diabetic gastroparesis treated with tegaserod over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females and males 18 to 75 years of age
* History of type I or type II diabetes mellitus for more than 3 years
* History of upper gastrointestinal symptoms consistent with diabetic gastroparesis
* Hemoglobin A1c < 9.5%
* Delayed gastric emptying

Exclusion Criteria:

* Abnormal endoscopy finding that can explain the presence of gastroparesis symptoms
* Medical conditions affecting gastric emptying
* A clinically significant medical condition that would interfere with the patient completing the trial
* Clinically significant abnormal creatinine level
* Known allergies to the same class of drug and/or allergies to eggs
* Severe obesity

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients treated with tegaserod that improve gastric emptying at Week 2 as compared with baseline via a solid phase technetium gastric emptying time (GET)

SECONDARY OUTCOMES:
Change from baseline in patients treated with tegaserod relative to: The proportion of patients that normalize gastric emptying
Symptoms of diabetic gastroparesis including postprandial fullness, early satiety, bloating, nausea and vomiting, and abdominal discomfort
Volume and symptomatic response to a gastric satiety drink test (GSDT)
Electrogastrography (EGG)
The safety and tolerability of tegaserod

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceutical Corporation, Study Chair — NPC
Locations (3):
- United States (3):
  - The University of Kansas Medical Center, Kansas City, Kansas
  - The University of Louisville, Louisville, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts